CLINICAL TRIAL: NCT04926168
Title: Randomized Pilot Study of Six Months Adjuvant Temozolomide (TMZ) vs No Adjuvant TMZ in Patients With Newly Diagnosed MGMT Methylated Glioblastoma (GBM) Following Standard Concurrent Radiation and TMZ
Brief Title: 6 Months Adjuvant Temozolomide (TMZ) vs No Adjuvant TMZ in Newly Diagnosed MGMT Methylated Glioblastoma (GBM)
Status: Withdrawn | Type: Observational
Why Stopped: lack of funds
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: ABTCv2-2101; IRB00285623 (Other: Johns Hopkins University)
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: MGMT-Methylated Glioblastoma
Keywords: TMZ; MGMT; adjuvant TMZ; GBM, Newly Diagnosed
MeSH Terms: conditions — Glioblastoma | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adjuvant TMZ (Treatment group):: Adjuvant TMZ (temozolomide) will be given to patients as standard of Care (SOC) treatment is administered on an outpatient basis.
  Patients will be provided with medication diaries and instructed in their use. TMZ will be dispensed as SOC.
  Interventions: Other: Standard of Care (SOC) Adjuvant TMZ (no intervention
- Delay TMZ (Observation group):: Patients in this cohort will have their TMZ in the adjuvant setting delayed and they will be observed with SOC procedures. Once the patient recurs, will be off "observation" and will be able to either have TMZ prescribed or something other.
  Interventions: Other: Delay of TMZ

INTERVENTIONS:
Other: Delay of TMZ — Delay of TMZ to analyze the current standard of care practice of prescribing TMZ post combination (RT and TMZ).
  Groups: Delay TMZ (Observation group):
Other: Standard of Care (SOC) Adjuvant TMZ (no intervention — SOC in Adjuvant Setting no intervention
  Groups: Adjuvant TMZ (Treatment group):

SUMMARY:
The primary objective of this trial is to evaluate overall survival of patients with O[6]-methylguanine-DNA methyltransferase (MGMT) methylated glioblastoma treated with or without six months of adjuvant TMZ after standard radiation (6000 centigray (cGy)) plus concurrent Temozolomide (TMZ).

Secondary Objectives include to prospectively assess the overall adverse event profile in the two treatment arms. To compare lymphocyte counts overtime between the two treatment arms and to prospectively compare quality of life in the two treatment arms as assessed by MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) and Neurological quality of Life/minimal infecting dose (NeuroQoL) (MID). The study will also compare progression-free survival between the two treatment arms.

DETAILED DESCRIPTION:
Recent phase III trials in patients with newly diagnosed patients with glioblastoma have demonstrated that adding new agents (such as cilengitide, bevacizumab, or nivolumab) to standard radiation and TMZ do not improve survival in this disease. The modest effects on survival observed with the Optune® device are offset by the high costs, inconvenience, and impact on the social interactions of patients wearing this device. Unfortunately, there are currently no novel therapies poised to displace the European Organization Research & Treatment Cancer (EORTC) regimen as the standard of care for patients with newly diagnosed Glioblastoma Multiforme (GBM).As a result, a formal evaluation of the efficacy of the 6 months of adjuvant TMZ in this regimen is important to patients and research studies.

This is of particular importance in the 40% of patients who have MGMT methylated glioblastoma. The very small benefit observed in MGMT unmethylated patients has led investigators in Europe and the United States of America (including Cancer Therapy Evaluation Program (CTEP) sponsored studies) to approve clinical trials in MGMT unmethylated patients with newly diagnosed glioblastoma that entirely omit TMZ in both the concurrent and the adjuvant settings Given the marginal value of TMZ in the MGMT unmethylated patient population, the investigator's propose to study the value of adjuvant TMZ in the subset of the MGMT methylated population. If omitting adjuvant TMZ is not detrimental to outcomes in the methylated population then it is extremely unlikely to benefit the unmethylated population where TMZ has even less effect.

Therefore, exploring the value of the six months of adjuvant TMZ in patients with newly diagnosed MGMT methylated glioblastoma is important. If this was shown to be of minimal value in prolonging survival there would be an immediate impact on both the standard care of patients and research efforts to improve therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patients must have a Karnofsky Performance Status ≥ 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
3. Patients must have had a pathologically confirmed recently diagnosed primary glioblastoma before they began concurrent radiation and temozolomide.
4. Patients must have tumor MGMT methylation status of methylated using a Clinical Laboratory Improvement Amendments (CLIA)-approved diagnostic test. Results of routinely-used methods for MGMT methylation testing (e.g. Mutagenically separated- polymerase chain reaction (MS-PCR) or quantitative PCR) are acceptable.
5. Documented mutated isocitrate dehydrogenase 1 gene (IDH1) isocitrate dehydrogenase 1 gene (IDH2)status: patients with either wild-type or(IDH) status are eligible. Patients with no documented status are also eligible and the status should be listed as unknown.
6. Patients must be completing or have completed 6 weeks of standard concurrent RT/TMZ.
7. Patients' post-operative treatment must have included at least 80% of standard radiation and concomitant temozolomide. Patients may not have received any other prior chemotherapy, immunotherapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes (TIL), lymphokine activated killer cells (LAK) or gene therapy), or hormonal therapy for their brain tumor. Prior Gliadel Wafers are allowed. Glucocorticoid therapy is allowed.
8. Patients must be clinically eligible for the six months of adjuvant temozolomide.
9. Patients must be able to provide written informed consent.
10. Patients must have baseline MRI performed within the 21 days prior to starting entering the "adjuvant" treatment or observation period.
11. Patients must have the following organ and marrow functions:

Absolute neutrophil count ≥1,500/µL Platelets ≥100,000/µL Hemoglobin ≥ 9 g/dL Total bilirubin ≤1.5 × institutional upper limit of normal (ULN), (except for patients with known Gilbert's syndrome who must have normal direct bilirubin) aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/ alanine transaminase (ALT) serum glutamic-pyruvic transaminase (SGPT) ≤ 2.5 × ULN Creatinine ≤1.5 × ULN OR Creatinine clearance ≥ 60 mL/min/1.73m2

Exclusion Criteria:

1. Patients receiving any other standard or investigational agents or who plan to use the OPTUNE device or other therapies for the glioblastoma are ineligible.
2. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible.
3. Patients must not have received prior RT, chemotherapy (except for their concurrent radiation and temozolomide for their recently diagnosed glioblastoma), immunotherapy or therapy with a biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes, lymphokine-activated killer cells, or gene therapy), or hormonal therapy for their brain tumor. Corticosteroid therapy is allowed.
4. Patients must not have had a prior diagnosis of a lower grade glioma.
5. No active treatment for other cancers in the past 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have completed 6weeks of TMZ + RT and have had good performance in that setting are eligible to be enrolled in this study to observe outcomes from being randomized to receive Standard of Care Adjuvant TMZ (6months TMZ 5 Days 1-5 or each cycle) or delay of adjuvant TMZ until recurrence post TMZ and RT. At recurrence patient may choose to start TMZ or some other treatment.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 2 years
  Compare overall survival with patients receiving adjuvant TMZ to those having TMZ delayed

SECONDARY OUTCOMES:
Grade 3 or above adverse events | 6 months
  Number of grade 3 or above adverse events
Change in Lymphocyte count | Up to 1 year
  Lymphocyte counts will be collected at baseline and every two months per standard care. Minimum measurements will be made three times through the course of trial, at baseline, 2 months from baseline measure, and a later measurement at 6 month or after. Linear mixed model will be carried out to compare the longitudinal profile of lymphocyte counts between the two arms.
Change in Quality of life as assessed by MDASI-BT | Up to 6 months
  A minimum of two reports are required for each patient, one at the baseline and another at time of first disease progression. Effort will be given to obtain the report at each standard clinical visit during the first 6 months (about 3 reports after enrollment). All MDASI-BT items are rated on numeric 0-to-10 scales, a low score indicates higher function.
Change in Quality of life as assessed by NeuroQoL/MID. | Up to 6 months
  A minimum of two reports are required for each patient, one at the baseline and another at time of first disease progression. Effort will be given to obtain the report at each standard clinical visit during the first 6 months (about 3 reports after enrollment). NeuroQoL/MID items are rated on numeric 0-to-10 scales, a low score indicates higher function.
Progression-free survival | Up to 2 years
  Time of progression-free survival is defined as date from randomization to date of progression as documented by treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Grossman, MD, Study Chair — Johns Hopkins University